CLINICAL TRIAL: NCT04811833
Title: Assessment of MonoPlus® Suture Material for Anastomosis in the Gastrointestinal Tract. A Prospective, Multi-centric, International, Single-arm, Observational Study in Daily Practice
Brief Title: Gastrointestinal Anastomosis Using MonoPlus® Suture
Acronym: GASTROMO
Status: Withdrawn | Type: Observational
Why Stopped: The GASTROMO study has been stopped early before enrolling its first patient because the results of our primary endpoint would have been inconsistent. The variability of the leakage rate between all anastomosis included in the study was overly high.
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2005
Record Dates: First submitted 2021-03-17; First posted 2021-03-23 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Gastrointestinal Stromal Tumors; Gastrointestinal Neoplasms; Digestive System Neoplasm; Stomach Tumor; Small Intestine Tumor; Colon Tumor; Rectum Tumor
Keywords: tumor disease; stomach tumor; small intestine tumor; colon tumor; rectum tumor; need for anastomosis
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Gastrointestinal Neoplasms; Digestive System Neoplasms; Stomach Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Monoplus®: Adult patients undergoing an elective, primary surgery within the gastrointestinal tract with the need for anastomosis.

SUMMARY:
The primary aim of this study is to collect clinical data on the performance of MonoPlus® suture applied in routine clinical practice. Diverse parameters are to be used to assess the safety and efficacy of MonoPlus® suture for gastrointestinal anastomosis construction.

This study has been designed to implement an action within the framework of a proactive Post Market Clinical Follow up (PMCF) activity.

ELIGIBILITY:
Inclusion criteria

* Adult patients undergoing an elective open or laparoscopic primary tumor resection within GI tract (stomach, small intestine, large intestine , colon and rectum.
* Age ≥ 18 years
* ASA ≤ III
* Written informed consent

Exclusion criteria

* ASA ≥IV
* Emergency operations
* Peritonitis
* Surgical interventions in the pancreas, oesophagus
* Patients with traumatic perforations
* Pregnant and/or breast-feeding women
* Patients who had received chemotherapy within the last 4 weeks or radiotherapy on the treated region within the last 2 weeks
* Patients who were receiving immunosuppressant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing an elective, primary surgery within the gastrointestinal tract with the need for ananastomosis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of anastomosis leakage rate at different timepoints in postoperative course | until 6 months after surgery
  The primary endpoint of this study is the anastomosis leakage rate until 6 months after surgery

SECONDARY OUTCOMES:
Comparison of dehiscence rate of the suture line at different timepoints in postoperative course | at discharge (approximately 10 days after surgery), 1 month and 6 months after surgery.
  Comparison of the dehiscence rate of the suture line at different postoperative examinations
Comparison of the Peritonitis rate at different timepoints in postoperative course | at discharge (approximately 10 days after surgery), 1 month, and 6 months after surgery
  Comparison of the Peritonitis rate of the suture line at different postoperative examinations
Comparison of the Surgical Site infection rate at different timepoints in postoperative course | at discharge (approximately 10 days after surgery), 1 month, and 6 months after surgery
  Incidence of postoperative surgical site infections, SSI (A1: Superficial incisional site infections and A2: Deep incisional surgical site infections) (efficacy parameter) Surgical Site Infection (SSI) is defined according to the definition of the US Centres for Disease Control and Prevention (CDC) at different postoperative examinations.
Comparison of bleeding at different timepoints in postoperative course | at discharge (approximately 10 days after surgery), 1 month, and 6 months after surgery
  Comparison of postoperative Bleeding rate at different postoperative examinations
Comparison of Abscess at different timepoints in postoperative course | at discharge (approximately 10 days after surgery), 1 month, and 6 months after surgery
  Comparison of postoperative Abscess rate at different postoperative examinations
Comparison of Postoperative Fistula at different timepoints in postoperative course | at discharge (approximately 10 days after surgery), 1 month, and 6 months after surgery
  Comparison of postoperative Fistula rate at different postoperative examinations
Comparison of Postoperative Perforation at different timepoints in postoperative course | at discharge (approximately 10 days after surgery), 1 month, and 6 months after surgery
  Comparison of postoperative Perforation rate at different postoperative examinations
Comparison of Postoperative Obstipation at different timepoints in postoperative course | at discharge (approximately 10 days after surgery), 1 month, and 6 months after surgery
  Comparison of postoperative Obstipation rate at different postoperative examinations
Comparison of Postoperative Stenosis at different timepoints in postoperative course | at discharge (approximately 10 days after surgery), 1 month, and 6 months after surgery
  Comparison of postoperative Stenosis rate at different postoperative examinations
Comparison of Reoperation rate due to an anastomosis leakage at different timepoints in postoperative course | at discharge (approximately 10 days after surgery), 1 month, and 6 months after surgery
  Comparison of Reoperation rate due to an anastomosis leakage at different postoperative examinations
Comparison of Mortality rate at different timepoints in postoperative course | at discharge (approximately 10 days after surgery), 1 month, and 6 months after surgery
  Comparison of postoperative Mortality rate at different postoperative examinations
Comparison of Stoma rate at different timepoints in postoperative course | at discharge (approximately 10 days after surgery), 1 month, and 6 months after surgery
  Comparison of postoperative Stoma rate at different postoperative examinations
Length of the overall postoperative hospital stay | until discharge (approximately 10 days postoperative)
  Number of days between date of surgery and date of discharge
Length of the postoperative stay in intensive care unit | until discharge (approximately 10 days postoperative)
  Number of days the patient has to stay in the intensive care unit after the intervention
Duration to perform the anastomosis | intraoperatively
  Time in Minutes the surgeon needs to perform the anastomosis
Course of Health Status | until 6 months postoperative
  EQ-5D-5L is a standardized measure of health status developed by EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. EQ-5D-5L is designed for self-completion by respondents and it takes only a few minutes to complete. Instructions to respondents are included in the questionnaire. EQ-5D-5L consists of 2 pages - descriptive system and the EQ visual Analogue scale (EQ-VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the respondents self rated health on a 20 cm vertical , visual analogue scale with endpoints labelled "the best health you can imagine" and " the worst health you can imagine"
Satisfaction of the patient with the surgery | at discharge (approximately 10 days postoperative), 1 month, and 6 months after surgery
  This parameter will be noted using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "maximal pain". The values are compared over postoperative period.
Assessment of suture material handling parameters | intraoperatively
  Assessment of the handling of the suture material intra-operatively using a questionnaire including different dimensions (knot security, tensile strength, knot run down, stiffness) with 5 evaluation levels (excellent, very good, good, satisfied, poor).

CONTACTS AND LOCATIONS:
Overall Officials: Wenceslao Vasquez Jimenez, Dr., Principal Investigator — Hospital General Universitario Gregorio Marañon
Locations (2):
- Spain (2):
  - Hospital Parc Taulí Sabadell, Sabadell, Catalonia
  - Servicio de Cirugía General y Digestiva, Sección cirugía, Madrid